CLINICAL TRIAL: NCT06196008
Title: SR2204: A Randomized Phase III Trial of a Perioperative Physical Activity Intervention in Older Adults With Lung Cancer and Their Family Caregivers
Brief Title: Telephone-based Physical Activity Coaching or Self Monitored Physical Activity to Improve Physical Function in Older Adults Who Are Undergoing Surgery for Lung Cancer and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23317; NCI-2023-09810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23317 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-01-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Telephone-based coaching session) (Experimental): Patients attend telephone-based coaching sessions over 20-50 minutes once 7-14 days before standard of care surgery, and then at days 7, 14, 21, and 51 post-discharge, for a total of 5 sessions. Patients also receive a personalized physical activity program and set fitness goals. FCGs also receive coaching and serve as a walking buddy for their patient. Patients and FCGs also wear an activity monitor throughout the trial.
  Interventions: Other: Educational Intervention; Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Written education) (Active Comparator): Patients receive written educational materials on physical activity and cancer survivorship. Patients and FCGs also wear an activity monitor throughout the trial.
  Interventions: Other: Educational Intervention; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend telephone-based coaching sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (Telephone-based coaching session)
Other: Educational Intervention — Receive written educational materials on physical activity and standard preoperative care
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (Written education)
Other: Exercise Intervention — Receive a personalized physical activity program, set fitness goals
  Arms: Arm I (Telephone-based coaching session)
Other: Medical Device Usage and Evaluation — Wear activity monitor
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares telephone-based physical activity coaching to self monitored physical activity for improving physical function in older adults who are undergoing surgery for lung cancer and their caregivers. Lung cancer surgery in older adults is associated with functional declines and unique challenges. Performing physical activity around the time of surgery has been shown to improve functional outcomes in patients and exercise programs delivered via telehealth may improve access and convenience for patients and minimize participant burden. Telephone-based physical activity coaching may improve physical functioning for older adults with lung cancer who are undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare changes from baseline in objective patient functional capacity as measured by 6 minute walk test (6MWT) at day 30 post-discharge between the two comparators.

SECONDARY OBJECTIVES:

I. To compare the following outcomes between the two comparators:

Ia. 6MWT at 60 and 180 days post discharge; Ib. Short Physical Performance Battery (SPPB) at 30, 60, and 180 days post-discharge; Ic. The following scores at 30, 60, and 180 days post-discharge: a) patient and family caregiver (FCG) reported self-efficacy; b) patient and FCG reported physical function; c) and patient and FCG quality of life (QOL); Id. Patient time at home and away from the hospital through 60 days post-discharge; Ie. Hospital readmissions rate and postoperative complications through 60 days post-discharge.

EXPLORATORY OBJECTIVES:

I. To explore associations between comparators, outcomes, and the following:

Ia. Perioperative, image-based sarcopenia using standard-of care preoperative chest computed tomography (CT) scans; Ib. Pedometer documented daily steps; Ic. Participant demographic and clinical characteristics.

OUTLINE: Patients and their FCG are randomized together to 1 of 2 arms.

ARM I: Patients attend telephone-based coaching sessions over 20-50 minutes once 7-14 days before standard of care surgery, and then at days 7, 14, 21, and 51 post-discharge, for a total of 5 sessions. Patients also receive a personalized physical activity program and set fitness goals. FCGs also receive coaching and serve as a walking buddy for their patient. Patients and FCGs also wear an activity monitor throughout the trial.

ARM II: Patients receive written educational materials on physical activity and cancer survivorship. Patients and FCGs also wear an activity monitor throughout the trial.

After completion of study intervention, patients are followed up at days 60 and 180 post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Documented informed consent of the participant and/or legally authorized representative
* PATIENT: Agreement to allow the use of preoperative chest CT scan for exploratory analysis, if available
* PATIENT: Agreement to wear pedometer during study duration

  * If unwilling, exceptions may be granted with study primary investigator (PI) approval
* PATIENT: Age >= 65 years
* PATIENT: Ability to read and understand English or Spanish and willingness to complete participant-reported outcomes and assessments
* PATIENT: Diagnosis of lung cancer or presumed lung cancer (as determined by surgeons) in patient
* PATIENT: Scheduled to undergo lung surgery for lung cancer or suspected lung cancer with curative intent (neoadjuvant therapy allowed)
* PATIENT: Adults lacking capacity to consent in the opinion of the attending surgeon will not be enrolled
* FCG: Documented informed consent of the participant and/or legally authorized representative
* FCG: Age >= 18
* FCG: Ability to read and understand English or Spanish and willingness to complete participant-reported outcomes and assessments
* FCG: Adults lacking capacity to consent in the opinion of the attending surgeon will not be enrolled

Exclusion Criteria:

* PATIENT: Lung surgery is scheduled in less than 14 calendar days from the time of registration
* PATIENT: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including exercise program and compliance issues related to feasibility/logistics)
* FCG: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including exercise program and compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2028-05-16 (Estimated); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Objective patient functional capacity | At 30 days post discharge
  Measured by the 6 minute walk test (6MWT). Analysis will be a study group comparison via linear regression model.

SECONDARY OUTCOMES:
Functional capacity | At 60 and 180 days post discharge
  Measured by 6MWT. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Lower extremity function | At 30, 60 and 180 days post discharge
  Measured by the short physical performance battery. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Patient and caregiver reported self efficacy | At 30, 60, and 180 days post discharge
  Measured by patient reported outcomes measurement information system (PROMIS) self efficacy. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Patient and caregiver reported physical function | At 30, 60 and 180 days post discharge
  Measured by PROMIS physical function. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Patient reported quality of life | At 30, 60 and 180 days post discharge
  Measured by Functional Assessment of Cancer Therapy -Lung for patients. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Caregiver reported quality of life | At 30, 60 and 180 days post discharge
  Measured by City of Hope-Quality of Life-Family Caregiver for caregivers. Will be assessed via repeated measures linear regression model with adjustment for baseline value of the outcome, stratification factors, and time point.
Patient time at home and away from the hospital | Up to 60 days post discharge
  Will be compared by study arm by linear regression models.
Hospital readmissions | Up to 60 days post discharge
  Will be compared by study arm via logistic regression.
Postoperative complications | Up to 60 days post discharge
  Will be compared by study arm via logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Raz, MD, Principal Investigator — City of Hope Medical Center
Locations (14):
- United States (13):
  - University of California, Davis, California
  - City of Hope Medical Center, Duarte, California
  - Standard University, Stanford, California
  - Yale New Haven Medical Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital (MGH) / Harvard, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- City of Hope at Georgia - Atlanta, Newnan, GA, Georgia

REFERENCES:
- [Derived] Sun V, Guthrie KA, Arnold KB, Antonoff M, Erhunmwunsee L, Borondy-Kitts A, Johnson J, Jones L, Ramirez M, Tong BC, Moremen JR, Yang CJ, Ng T, Kim SS, Brown LM, Blasberg JD, Lui NS, Kneuertz PJ, Toloza EM, Kim JY, Raz DJ. Comparative effectiveness of perioperative physical activity in older adults with lung cancer and their family caregivers: design of a multicenter pragmatic randomized trial. BMC Cancer. 2024 Aug 8;24(1):976. doi: 10.1186/s12885-024-12660-5. PMID 39118035